CLINICAL TRIAL: NCT03334487
Title: Open-Label, Single Arm, Phase 3b Study Evaluating the Safety of Rovalpituzumab Tesirine for Third-Line and Later Treatment of Subjects With Relapsed or Refractory DLL3 Expressing Small Cell Lung Cancer
Brief Title: Study Evaluating the Safety of Rovalpituzumab Tesirine for Third-Line and Later Treatment of Subjects With Relapsed or Refractory Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-292; 2017-003173-33 (EudraCT Number)
Expanded Access: NCT03503890 (No longer available)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Small Cell Lung Cancer
Keywords: Cancer; Small Cell Lung Cancer; Relapsed Small Cell Lung Cancer; Remitting Small Cell Lung Cancer; Delta-like protein 3 (DLL3); DLL3 Expressing Small Cell Lung Cancer; Rovalpituzumab Tesirine
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Dexamethasone; rovalpituzumab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rovalpituzumab tesirine + dexamethasone (Experimental): Rovalpituzumab tesirine 0.3 mg/kg administered intravenously on Day 1 of each 6-week cycle plus oral dexamethasone 8 mg twice daily on Day -1, Day 1, and Day 2 of 6-week each cycle.
  Interventions: Drug: Dexamethasone; Drug: Rovalpituzumab tesirine

INTERVENTIONS:
Drug: Dexamethasone — Oral
Drug: Rovalpituzumab tesirine — Intravenous
  Other Names: SC16LD6.5

SUMMARY:
A single-arm, open-label study to assess the overall safety of rovalpituzumab tesirine in participants with relapsed or refractory delta-like protein 3 (DLL3) expressing small cell lung cancer by evaluating the frequency of high grade (>= Grade 3) select treatment-emergent adverse events (TEAEs).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Minimum life expectancy of at least 12 weeks.
* Laboratory values meeting the criteria specified in the protocol.
* Histologically or cytologically confirmed Small Cell Lung Cancer (SCLC) with documented disease progression after at least 2 prior systemic regimens, including at least one platinum-based regimen.
* Delta-Like Protein 3 (DLL3)-expressing SCLC based on central immunohistochemistry (IHC) assessment of banked or otherwise representative tumor tissue.
* Measurable disease as described per protocol.
* In participants with a history of central nervous system (CNS) metastases, documentation of stable or improved status based on brain imaging for at least 2 weeks after completion of definitive treatment and within 2 weeks prior to first dose of study drug, off or on a stable dose of corticosteroids.

Exclusion Criteria:

* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association Class III - IV within 6 months prior to first dose of study drug.
* Recent or on-going serious infection.
* History of other invasive malignancy that has not been in remission for at least 3 years.
* History of exposure to a pyrrolobenzodiazepine (PBD)-based drug or known hypersensitivity to rovalpituzumab tesirine or excipient contained in the drug formulation.
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells.
* Documented history of capillary leak syndrome.
* Grade 2 or higher pleural or pericardial effusion within 4 weeks of investigational drug start, or earlier history of recurrent Grade 2 or higher effusions with ongoing requirements for pericardiocentesis or thoracentesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a High Grade (>= Grade 3) Protocol Specified TEAE | Approximately 32 months
  Number of participants with a high grade (≥ Grade 3) protocol specified Treatment-Emergent Adverse Events (TEAEs) during and after treatment with rovalpituzumab tesirine. Severity of TEAEs will be graded at each study visit according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03.

SECONDARY OUTCOMES:
Change in Participant Reported Outcome EORTC QLQC15-PAL | Approximately 32 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Palliative Cancer (EORTC QLQ-C15-PAL) is a 15-item self-report questionnaire composed of 4 multi-item scales (physical & emotional functioning, fatigue and pain) along with 6 individual items (nausea & vomiting, dyspnea, insomnia, appetite loss, constipation, and global quality of life).
Progression Free Survival (PFS) | Approximately 32 months
  PFS is based on independent review of radiographic assessment, defined as the time from randomization to documented disease progression or death from any cause, whichever occurs earlier.
Overall Survival (OS) | Approximately 32 months
  Overall Survival (OS) is defined as the time from the date of randomization to the date of death from any cause.
Objective response rate (ORR) | Approximately 32 months
  ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Change in EORTC QLQ-LC-13 | Approximately 32 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer (EORTC QLQ-LC 13) is a lung cancer specific module developed to assess lung cancer-associated symptoms and treatment-related side effects among lung cancer patients.
Duration of Objective Response (DOR) | Approximately 32 months
  DOR is defined as the time between the date of first response (CR or PR, whichever is recorded first) to the date of the first documented tumor progression (per RECIST version 1.1) or death due to any cause, whichever comes first.
Clinical Benefit Rate (CBR) | Approximately 32 months
  CBR is defined as the proportion of participants with an objective response or stable disease (CR+PR+SD) according to RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (60):
- United States (27):
  - Ironwood Cancer & Res Ctr /ID# 171335, Chandler, Arizona
  - Mayo Clinic - Scottsdale /ID# 171359, Scottsdale, Arizona
  - VA Central California Health C /ID# 170951, Fresno, California
  - Loma Linda University Medical /ID# 171377, Loma Linda, California
  - UC Irvine Health /ID# 171343, Orange, California
  - Kaiser Permanente - Roseville /ID# 200779, Roseville, California
  - Kaiser Permanente-Santa Clara /ID# 203024, Santa Clara, California
  - Kaiser Permanente Medical Ctr-Vallejo /ID# 169758, Vallejo, California
  - Kaiser Permanente- Walnut Creek /ID# 201305, Walnut Creek, California
  - Univ of Colorado Cancer Center /ID# 200810, Aurora, Colorado
  - Boca Raton Regional Hospital /ID# 200168, Boca Raton, Florida
  - UMHC/Sylvester Comprehensive /ID# 171462, Deerfield Beach, Florida
  - Mount Sinai Comp Cancer Ctr /ID# 169759, Miami, Florida
  - Illinois Cancer Care, PC /ID# 171310, Peoria, Illinois
  - Baptist Health /ID# 171379, Lexington, Kentucky
  - Norton Cancer Institute /ID# 200827, Louisville, Kentucky
  - Tulane Cancer Center Clinic /ID# 171376, New Orleans, Louisiana
  - Sandra Malcolm Berman Cncr Ins /ID# 171346, Baltimore, Maryland
  - St. Luke's University Hospital /ID# 171374, Duluth, Minnesota
  - Valley Hospital - Westwood, NJ /ID# 171357, Westwood, New Jersey
  - Wake Forest Baptist Medical Center /ID# 169799, Winston-Salem, North Carolina
  - The Ohio State University Comp /ID# 171352, Columbus, Ohio
  - St. Luke's Hematology Oncology /ID# 171378, Bethlehem, Pennsylvania
  - Tennessee Oncology PLLC: Sarah /ID# 171380, Nashville, Tennessee
  - Vanderbilt Ingram Henry Cancer /ID# 171356, Nashville, Tennessee
  - VCS, Virginia Cancer Specialis /ID# 169760, Arlington, Virginia
  - Kadlec Clinic Hematology and O /ID# 169797, Kennewick, Washington
- Australia (6):
  - Coffs Harbour Health Campus /ID# 200642, Coffs Harbour, New South Wales
  - The Tweed Hospital /ID# 200646, Tweed Heads, New South Wales
  - The Townsville Hospital /ID# 200640, Douglas, Queensland
  - Austin Hospital /ID# 200639, Heidelberg, Victoria
  - Border Medical /ID# 200645, Wodonga, Victoria
  - Perron Institute for Neurological and Translational Science /ID# 200644, Nedlands, Western Australia
- Brazil (8):
  - Bahia Oncology Center - NOB /ID# 201272, Salvador, Estado de Bahia
  - Associação Hospital de Caridade Ijuí - Centro de Tratamento de Cancer - CACON /ID# 200496, Ijuí, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS /ID# 201258, Porto Alegre, Rio Grande do Sul
  - Icesp /Id# 201036, São Paulo, São Paulo
  - Inca /Id# 202594, Rio de Janeiro
  - Instituto COI de Educacao e Pe /ID# 200499, Rio de Janeiro
  - Fundacao Antonio Prudente /ID# 200218, São Paulo
  - Hospital de Cancer de Barretos /ID# 200104, São Paulo
- Canada (4):
  - Tom Baker Cancer Centre /ID# 171561, Calgary, Alberta
  - QE II Health Sciences Centre /ID# 171569, Halifax, Nova Scotia
  - London Health Sciences Centre /ID# 171567, London, Ontario
  - The Ottawa Hospital /ID# 200682, Ottawa, Ontario
- Germany (7):
  - Franziskus-Hospital Harderberg /ID# 201145, Georgsmarienhütte, Lower Saxony
  - Charite Universitatsmedizin B- /ID# 170079, Berlin
  - Asklepios Fachkliniken M. Gaut /ID# 170081, Gauting
  - Thoraxklinik Heidelberg gGmbH /ID# 170078, Heidelberg
  - Klinikum Kassel - Onkologie /ID# 170083, Kassel
  - Universitatsklinikum Munster /ID# 170087, Münster
  - Pius Hospital Oldenburg /ID# 170080, Oldenburg
- Sweden (5):
  - Akademiska Sjukhuset /ID# 171248, Uppsala, Uppsala County
  - Gavle Hospital /ID# 171253, Gävle
  - University Hospital Linkoping /ID# 201666, Linköping
  - Karolinska University Hospital /ID# 201967, Stockholm
  - Norrlands Universitetssjukhus /ID# 171250, Umeå
- United Kingdom (3):
  - Leicester Royal Infirmary /ID# 201154, Leicester, England
  - Christie NHS Foundation Trust /ID# 201149, Manchester
  - Royal Preston Hospital /ID# 201146, Preston

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html